CLINICAL TRIAL: NCT03807544
Title: Study to Optimize and Validate the Treatment Parameters for the Empower Neuromodulation System
Brief Title: Treatment Parameters for the Empower Neuromodulation System (ENS)
Acronym: AUD1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD-12-1154
Record Dates: First submitted 2019-01-04; First posted 2019-01-17 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Use Disorder
Keywords: AUD; TENS
MeSH Terms: conditions — Alcoholism | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- TENS treatment arm (Experimental): This study is a usability study, where all subjects will receive the same experimental treatment for their single visit.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — Transcutaneous electrical nerve stimulation

SUMMARY:
The subject will be administered a treatment at a treatment location and then be asked if he/she believes it is the active treatment, sham treatment, or does not know. A clinical-grade nerve conduction assessment system will be used both to provide electrical stimulation at four locations to record peripheral responses. The subject will self-administer two treatment sessions at two active treatment sites.

ELIGIBILITY:
Inclusion Criteria:

1. Is 21-75 years old
2. Can provide informed consent
3. Currently has a stable living situation
4. Had one heavy drinking week (>7 drinks/week for women; >14 drinks/week for men) over the past 6 months
5. Has a breath alcohol concentration of 0.00% at enrollment
6. Is willing to follow all study procedures

Exclusion Criteria:

1. Has been diagnosed with schizophrenia, epilepsy, peripheral neuropathy, or nerve damage
2. Has implanted electrical and/or neurostimulator device (e.g. pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, sacral stimulator, bone growth stimulator, or cochlear implant)
3. Has a tattoo or conductive, ferromagnetic, or other magnetic-sensitive metals that cannot be removed from the hand, wrist, or biceps
4. Is currently pregnant or breastfeeding
5. Has a bleeding disorder, a history of deep vein thrombosis, or is on anticoagulation drugs
6. Has used an investigational drug/device therapy within the past 4 weeks
7. Is deemed unsuitable for enrollment in study by the PI

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TheraNova, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TENS Treatment Arm: This study is a usability study, where all subjects will receive the same experimental treatment (both palms and wrists) for their single visit. TENS: Transcutaneous electrical nerve stimulation
Period: Overall Study
Arm/Group | TENS Treatment Arm
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy adults
Arm/Group | TENS Treatment Arm
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: Years] | 46.82 [23 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Effective Electrode Placement
Description: Compare two active treatment electrode locations to evaluate the effect of electrode placement on the appearance of sensory nerve action potentials, including tingling sensation, along the stimulated nerve using electromyography (EMG).
Time Frame: 2 hours, length of study visit
Measure: Count of Participants; unit: Participants
Groups:
- TENS Location - Palm: Measuring SNAP/Tingling off of the Palm location (active treatment site)
- TENS Location - Wrist: Measuring SNAP/Tingling off of the Wrist location (active treatment site)
Arm/Group | TENS Location - Palm | TENS Location - Wrist
Number analyzed (Participants) | 17 | 17
Participants | 17 | 17

ADVERSE EVENTS:
Time Frame: One 2-hour visit
Arm/Group | TENS Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT03807544/Prot_SAP_000.pdf